CLINICAL TRIAL: NCT03598270
Title: A Phase III Randomized, Double-blinded Trial of Platinum-based Chemotherapy With or Without Atezolizumab Followed by Niraparib Maintenance With or Without Atezolizumab in Patients With Recurrent Ovarian, Tubal or Peritoneal Cancer and Platinum Treatment-free Interval (TFIp) >6 Months
Brief Title: Platinum-based Chemotherapy With Atezolizumab and Niraparib in Patients With Recurrent Ovarian Cancer
Acronym: ANITA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: Hoffmann-La Roche (Industry); GlaxoSmithKline (Industry); AGO Study Group (Other); Belgian Gynaecological Oncology Group (Other); ARCAGY/ GINECO GROUP (Other); Israeli Society of Gynecologic Oncology (Other); MaNGO (Unknown); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENGOT-Ov41/GEICO 69-O/ANITA; 2018-000366-11 (EudraCT Number); ENGOT-Ov41 (Other: ENGOT); GEICO 69-O (Other: GEICO)
Record Dates: First submitted 2018-06-02; First posted 2018-07-26 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Ovarian Carcinoma
Keywords: Ovarian; Atezolizumab; Niraparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel; niraparib; Gemcitabine; liposomal doxorubicin; atezolizumab

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, multi-center study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Atezolizumab and placebo treatment will be double blinded, unknown to both the subject and the study staff, including the treating physician. In order to maintain the blind, atezolizumab and placebo will be identical in appearance and packaging.
  The study medication will be labeled using a unique kit id number, which is linked to the randomization scheme. The active and placebo kits will be presented in the same packaging to ensure blinding of the study medication Individual treatment codes, indicating the treatment randomization for each randomized patient, will be available to the investigator(s) or pharmacists from the IVRS/IWRS. Routines for this will be described in the Interactive Voice Response System/Interactive Web Response System (IVRS/IWRS) user manual that will be provided to each centre.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Control Arm) (Placebo Comparator): Placebo of atezolizumab in combination with one of the platinum based regimens below (investigator's choice) followed by maintenance niraparib with placebo:
  * Carboplatin (AUC = 5, d1) plus paclitaxel and placebo every 3 weeks. Non-progressing patients will be switched to maintenance niraparib in combination with placebo every 3 weeks
  * Carboplatin (AUC = 4, d1) plus gemcitabine and placebo every 3 weeks. Non-progressing patients will be switched to maintenance niraparib in combination with placebo every 3 weeks.
  * Carboplatin (AUC = 5, d1) plus pegylated liposomal doxorubicin (PLD) and placebo every 4 weeks. Non-progressing patients will be switched to maintenance niraparib in combination with placebo every 3 weeks.
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Paclitaxel; Drug: Niraparib; Drug: Gemcitabine; Drug: Pegylated liposomal doxorubicin (PLD)
- Arm B (experimental arm) (Experimental): Atezolizumab in combination with one of the platinum based regimens below (investigator's choice) followed by maintenance niraparib with atezolizumab:
  * Carboplatin (AUC = 5, d1) plus paclitaxel and atezolizumab every 3 weeks. Non-progressing patients will be switched to maintenance niraparib in combination with atezolizumab every 3 weeks.
  * Carboplatin (AUC = 4, d1) plus gemcitabine and atezolizumab every 3 weeks. Non-progressing patients will be switched to maintenance niraparib in combination with atezolizumab every 3 weeks.
  * Carboplatin (AUC = 5, d1) plus pegylated liposomal doxorubicin (PLD) and atezolizumab every 4 weeks. Non-progressing patients will be switched to maintenance niraparib in combination with atezolizumab every 3 weeks.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Niraparib; Drug: Gemcitabine; Drug: Pegylated liposomal doxorubicin (PLD); Drug: Atezolizumab

INTERVENTIONS:
Drug: Placebo — Volume equivalent to 1200 mg of atezolizumab drug product. Intravenous Day 1
  Other Names: Placebo of Atezolizumab
  Arms: Arm A (Control Arm)
Drug: Carboplatin — Intravenous. Day 1
Drug: Paclitaxel — 175 mg/m². Intravenous. Day 1
Drug: Niraparib — 200 mg or 300 mg. Oral. From day 1 to 21
Drug: Gemcitabine — 1000 mg/m². Intravenous. Day 1 and day 8.
Drug: Pegylated liposomal doxorubicin (PLD) — 30 mg/m². Intravenous. Day 1
Drug: Atezolizumab — 1200 mg. Intravenous. Day 1
  Other Names: Tecentriq
  Arms: Arm B (experimental arm)

SUMMARY:
Atezolizumab in this study is expected to have a positive benefit-risk profile for the treatment of patients with platinum-sensitive relapse of ovarian cancer. Of interest, atezolizumab is being investigated also in combination with platinum-based doublet chemotherapy in second line (2L)/ third line (3L) platinum-sensitive recurrent ovarian cancer patients in ATALANTE (NCT02891824), which also includes bevacizumab in the combination. The study is proceeding as expected after >100 patients enrolled and under independent Data Monitoring Committee (IDMC) supervision.

Platinum-containing therapy is considered the treatment of choice for patients with platinum-sensitive relapse. However the duration of response and the prolongation of the progression free interval with chemotherapy are usually brief, among other because these chemotherapy regimens cannot be continued until progression as they are associated with neurological, renal and hematological toxicity and cannot generally be tolerated for more than about 6 to 9 cycles.

Niraparib received FDA approval in March 2017 as maintenance treatment of adult patients with recurrent epithelial ovarian, fallopian tube or primary peritoneal cancer who are in complete or partial response to platinum-based chemotherapy. Recently, the European Medicines Agency (EMA) has also approved niraparib as maintenance monotherapy. Despite the progress brought about by niraparib, there is a need for a more effective treatment to extend the progression free interval in this patient population. The combination with immune checkpoint inhibitors such as anti-death protein 1 (anti-PD1) or anti-death protein ligand 1 (anti-PD-L1) has a compelling rationale to this aim, especially under the light of the emerging clinical data of this combination.

The use of atezolizumab concurrent to platinum-containing chemotherapy followed by niraparib as maintenance therapy after completion of chemotherapy, as per normal clinical practice, may provide further benefit to patients in terms of prolonging the progression free interval and increasing the interval between lines of chemotherapy, hence delaying further hospitalization and the cumulative toxicities associated with chemotherapy. Additionally, preliminary studies with atezolizumab suggest an acceptable tolerability profile for long term clinical use in recurrent ovarian cancer patients and other indications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Life expectancy ≥3 months
3. Signed informed consent and ability to comply with treatment and follow-up
4. Histologically confirmed diagnosis (cytology alone excluded) of high- grade serous or endometrioid ovarian, primary peritoneal or tubal carcinoma.
5. Breast Cancer (BRCA) mutational status is known (germline or somatic)
6. Relapsed disease more than 6 months after the last platinum dose
7. No more than 2 prior lines of chemotherapy are allowed, and the last one must contain a platinum-based regimen
8. At least one measurable lesion to assess response by RECIST v1.1 criteria.
9. Mandatory de novo tumor biopsy (collected within 3 months prior to randomization) sent to HistoGene X as a formalin-fixed, paraffin-embedded (FFPE) sample for PD-L1 status determination for randomization. The inclusion of patients with non informative tissue PD-L1 status will be capped to 10% of the whole study population:

   * If the mandatory de novo biopsy is technically not possible or failed to produce enough representative tumor tissue, an FFPE sample from archival tissue may be acceptable after approval of the sponsor.
   * Bone metastases, fine needle aspiration, brushing, cCell pellet from pleural effusion, or ascites or lavage are not acceptable.
10. Two additional tumour samples are needed: Archival tumor sample must be available for exploratory PD-L1 testing in archival tissue and archival or "de novo" tissue sample for biomarkers must also be available.
11. Performance status determined by Eastern Cooperative Oncology Group (ECOG) score of 0-1
12. Normal organ and bone marrow function:

    * Haemoglobin ≥10.0 g/dL
    * Absolute neutrophil count (ANC) ≥1.5 x 109/L
    * Lymphocyte count ≥0.5 × 109/L
    * Platelet count ≥100 x 109/L
    * Total bilirubin ≤1.5 x institutional upper limit of normal (ULN)
    * Serum albumin ≥2.5 g/dL
    * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5 x ULN, unless liver metastases are present in which case they must be ≤5 x ULN
    * Serum creatinine ≤1.5 x institutional ULN or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
    * Patients not receiving anticoagulant medication must have an International Normalized Ratio (INR) ≤1.5 and an Activated ProThrombin Time (aPTT) ≤1.5 x ULN.
13. Negative Test Results for Hepatitis.
14. Toxicities related to previous treatments must be recovered to < grade 2
15. Female participants must be postmenopausal or surgically sterile or otherwise have a negative serum pregnancy test within 7 days of the first study treatment and agree to abstain from heterosexual intercourse or use single or combined contraceptive methods.
16. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
17. Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.

Exclusion Criteria:

1. Non-epithelial tumor of the ovary, the fallopian tube or the peritoneum.
2. Ovarian tumors of low malignant potential or low grade
3. Other malignancy within the last 5 years except curatively treated non-melanoma skin cancer, in situ cancer of the cervix and ductal carcinoma in situ (DCIS)
4. Major surgery within 4 weeks of starting study treatment or patients who have not completely recovered (Grade ≥ 2) from the effects of any major surgery at randomization
5. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1, Cycle 1
6. Administration of other chemotherapy drugs, anticancer therapy or anti-neoplastic hormonal therapy, or treatment with other investigational agents or devices within 28 days prior to randomization, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, or anticipation to do it during the trial treatment period (non-investigational hormonal replacement therapy is permitted)
7. Palliative radiotherapy (e.g., for pain or bleeding) within 6 weeks prior to randomization or patients who have not completely recovered (Grade ≥ 2) from the effects of previous radiotherapy
8. Current or recent (within 10 days prior to randomization) chronic use of aspirin (>325 mg/day) or clopidogrel (>75 mg/day)
9. Clinically significant (e.g. active) cardiovascular disease
10. Resting ECG with corrected QT interval (QTc) >470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
11. Left ventricular ejection fraction defined by multigated acquisition/echocardiogram (MUGA/ECHO) below the institutional lower limit of normal
12. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to randomization) in case of suspected spinal cord compression
13. History or evidence upon neurological examination of central nervous system (CNS) disorders (e.g. uncontrolled epileptic seizures) unless adequately treated with standard medical therapy
14. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease
15. Uncontrolled tumor-related pain
16. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed
17. Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium or calcium >12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
18. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications
19. Pregnant or lactating women
20. Simultaneously receiving therapy in any interventional clinical trial
21. Prior treatment with CD137 agonists or immune checkpoint stimulating or blockade therapies, such as anti-PD1, anti-PDL1 or anti-CTLA4 therapeutic antibodies
22. Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha (IFN-α) and interleukin-2 (IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
23. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF) agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial
24. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
25. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis
26. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
27. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
28. Active tuberculosis
29. Administration of a live, attenuated vaccine (including against influenza) within 4 weeks prior to Cycle 1, Day 1 or anticipation that it will be administered at any time during the treatment period of the study or within 5 months after the final dose of atezolizumab.
30. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
31. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation or allergy to any of the other drugs included in the protocol or their solvents (including to Cremophor®)
32. Patient has received prior treatment with a poly (adenosine diphosphate (ADP)-ribose) polymerase (PARP) inhibitor in the recurrent setting or has participated in a study where any treatment arm included administration of a PARP inhibitor in the recurrent setting, unless the patient is unblinded and there is evidence of not having received a PARP inhibitor. Patients that received PARP inhibitor as front line are eligible for the study. The duration of exposure to PARPi following front line therapy needs to be ≥18 months for BRCA mutated patients and ≥ 12 months for BRCA wild type patients.
33. Patient has had any known ≥Grade 3 hematological toxicity anemia, neutropenia or thrombocytopenia due to prior cancer chemotherapy that persisted >4 weeks and was related to the most recent treatment
34. Patient has any known history or current diagnosis of Myelodysplasic syndrome (MDS) or Anaplastic Myeloid Leukemia (AML)
35. Previous allogeneic bone marrow transplant or previous solid organ transplantation
36. Patient has a condition (such as transfusion dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results or interfere with the patient's participation for the full duration of the study treatment
37. Participant has any known hypersensitivity to niraparib components or excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 417 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 30 months
  Period from study entry (day of randomization) until disease progression, death or date of last contact. Progression will be based on tumor assessment made by the investigators according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | 60 months
  The observed length of life from entry into the study (day of randomization) to death due to any cause, or the date of last contact if patient alive.
Time to first subsequent therapy or death (TFST) | 60 months
  Time from the date of randomization in the current study to the start date of the first subsequent anticancer therapy.
Time to second subsequent therapy or death (TSST) | 60 months
  Time from the date of randomization in the current study to the start date of the second subsequent anticancer therapy
Time to second progression or death (PFS2) | 60 months
  Time from treatment randomization to the earliest date of assessment of progression on the next anticancer therapy following study treatment or death by any cause.
Incidence of Treatment Adverse Events | 60 months
  Frequency and severity of adverse events as assessed by CTCAE version 5.0 for the regimens administered on this study
Patient-reported abdominal symptoms | 60 months
  Clinically-meaningful improvement in patient-reported abdominal pain or bloating, defined as a 10-point decrease from the baseline score on either of the two items of the EORTC quality of life questionnaire-ovarian cancer module (QLQ-OV28) abdominal/GI symptom scale (items 31 and 32)
Patient-reported outcomes (PROs) of function and health related quality of life (HRQoL) | 60 months
  Clinical improvement, remaining stable, or deterioration in patient-reported function and HRQoL, defined as a 10-point increase, changes within 10 points, and a 10-point decrease, respectively, from the baseline score on each of the functional (physical, role, emotional, and social) and global health status/HRQoL scales of EORTC QLQ-C30
Objective Response Rate (ORR) | 60 months
  Based on investigator assessment by RECIST v1.1 during the chemotherapy phase and during the maintenance phase
Duration of response (DOR) | 60 months
  Based on investigator assessment by RECIST v1.1 during the chemotherapy phase and during the maintenance phase
Progression-free survival (PFS) from the beginning of the maintenance phase in all patients, in patients in complete or partial response after completing chemotherapy and in patients with stable disease after completing chemotherapy | 60 months
  Period from start of maintenance treatment until disease progression, death or date of last contact assessed by the investigator according to RECIST v1.1 criteria, in all patients receiving maintenance treatment as well as in the subgroup of patients with complete response/partial response (CR/PR) of stable disease (SD) after completing chemotherapy
Progression Free Survival (PFS) and BRCA status. | 60 months
  Relationship of PFS with BRCA mutational status
Overall Survival (OS) and BRCA status. | 60 months
  Relationship of OS with BRCA mutational status
Time to first subsequent therapy or death (TFST) and BRCA status. | 60 months
  Relationship of TFST with BRCA mutational status
Objective Response Rate (ORR) and BRCA status. | 60 months
  Relationship of ORR with BRCA mutational status
Duration of Response (DOR) and BRCA status. | 60 months
  Relationship of DOR with BRCA mutational status
Progression Free Survival (PFS) and PD-L1 status | 60 months
  Relationship of PFS with PD-L1 expression status
Overall Survival (OS) and PD-L1 status | 60 months
  Relationship of OS with PD-L1 expression status
Time to first subsequent therapy or death (TFST) and PD-L1 status | 60 months
  Relationship of TFST with PD-L1 expression status
Objective Response Rate (ORR) and PD-L1 status | 60 months
  Relationship of ORR with PD-L1 expression status
Duration of Response (DOR) and PD-L1 status | 60 months
  Relationship of DOR with PD-L1 expression status
Efficacy of atezolizumab compared to placebo in the PD-L1 negative and PD-L1 positive subgroups | 60 months
  To evaluate the immune response to atezolizumab

OTHER OUTCOMES:
Evaluate PROs of disease associated with atezolizumab versus placebo | 60 months
  Mean and mean changes from the baseline score in disease by cycle and between treatment arms as assessed by scale of european organization for research and treatment of cancer quality of life questionnaire core-30 (EORTC QLQ-C30)
Evaluate PROs of disease associated with atezolizumab versus placebo | 60 months
  Mean and mean changes from the baseline score in disease by cycle and between treatment arms as assessed by scale quality of life questionnaire ovarian 28 (QLQ-OV28)
Evaluate treatment-related symptoms associated with atezolizumab versus placebo | 60 months
  Mean and mean changes from the baseline score in treatment-related symptoms by cycle and between treatment arms as assessed by all symptom item scale of EORTC QLQ-C30.
Evaluate treatment-related symptoms associated with atezolizumab versus placebo | 60 months
  Mean and mean changes from the baseline score in treatment-related symptoms by cycle and between treatment arms as assessed by all symptom item scale of EORTC QLQ-OV28
Treatment burden | 60 months
  Any treatment burden patients may experience in association with atezolizumab versus placebo, as measured by a single item (from GP5: "I am bothered by side effects of treatment") from the physical wellbeing subscale of the Functional Assessment of Cancer Therapy - General (FACT-G) Quality of Life instrument
Patients' health utility | 60 months
  Evaluate and compare between treatment arms patients' health utility as measured by European Quality of Life Visual Analogue Scale (EQ-VAS) to generate utility scores for use in economic models for reimbursement
Patients' health utility | 60 months
  Evaluate and compare between treatment arms patients' health utility as measured by EuroQoL 5 Dimension to generate utility scores for use in economic models for reimbursement
Patients' health utility | 60 months
  Evaluate and compare between treatment arms patients' health utility as measured by 5 Level Questionnaire (EQ-5D-5L) to generate utility scores for use in economic models for reimbursement
Association of PD-L1 expression and other immune biomarkers with clinical outcomes | 60 months
  Relationship between tumour immune-related or disease type-related biomarkers (including but not limited to mutational burden, PD-L1, tumor-infiltrating lymphocytes (TILs) and cluster of differentiation (CD)8) in tumour tissues or blood samples, and clinical outcomes
Biomarkers predictive of the response to atezolizumab. | 60 months
  Relationship between exploratory biomarkers (circulating cell-free DNA) assessed from plasma before and during/after treatment, and clinical outcomes
Biomarkers predictive of the response to atezolizumab. | 60 months
  Relationship between exploratory biomarkers (proteins) assessed from plasma before and during/after treatment, and clinical outcomes
Biomarkers predictive of the response to atezolizumab. | 60 months
  Relationship between exploratory biomarkers (cytokines) assessed from plasma before and during/after treatment, and clinical outcomes
Effect of antibiotic (ATB) use on the efficacy of atezolizumab. | 60 months
  Relationship between ATB use within 2 month before and 1 month after the first study administration with atezolizumab efficacy as measured by PFS.
To evaluate the efficacy of atezolizumab vs placebo according to previous use of PARP inhibitors in front line. | 60 months
  Relationship between previous use of PARP inhibitors in front line and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio González Martín, MD PhD, Principal Investigator — Clinica Universitaria de Navarra
Locations (71):
- Belgium (5):
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Leuven, Leuven
  - CHU de Liège, site Sart Tilman, Liège
  - CHU Ambroise Paré, Mons
  - CHU UCL Namur site St. Elisabeth, Namur
- France (20):
  - ICO - Paul Paupin - ANGERS, Angers
  - CHU Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - ONCOGARD - Institut de Cancérologie du Gard, Nîmes
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Diaconesses-Croix Saint Simon, Paris
  - Hôpital Tenon, Paris
  - HPCA Cario, Plérin
  - Institut Curie - Hopital Claudius Régaud, Saint-Cloud
  - Institut Curie - Hôpital René Huguenin- SAINT CLOUD, Saint-Cloud
  - ICO Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (14):
  - Hochtaunus-Kliniken, Bad Homburg
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Kliniken Essen-Mitte, Essen
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Diakovere Krankenhaus, Hanover
  - Klinikum Kulmbach, Kulmbach
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Münster, Münster
  - MVZ Nordhausen, Nordhausen
  - Klinikum Oldenburg AöR, Oldenburg
  - ROMed Klinikum Rosenheim, Rosenheim
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsfrauenklinik Ulm, Ulm
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
- Italy (7):
  - Spedali Civili, Brescia
  - Asst Lecco, Lecco
  - Istituto Europeo di Oncologia, Milan
  - I.R.C.C.S. Istituto Oncologico Veneto, Padua
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - AO Città della Salute e della Scienza- Ospedale Sant'Anna, Torino
  - Ospedale Mauriziano Umberto I, Torino
- Spain (25):
  - Hospital de Sabadell, Sabadell, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de A Coruña, A Coruña
  - ICO Badalona, Badalona
  - H. Clínic Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de la Vall d'Hebron, Barcelona
  - H Reina Sofía Cordoba, Córdoba
  - ICO Girona, Girona
  - ICO Hospitalet, Hospitalet Del Llobregat
  - Hospital de León, León
  - Clinica Universitaria de Navarra, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Complejo Hospitalario Regional de Málaga, Málaga
  - H Morales Meseguer, Murcia
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Virgen del Rocio, Seville
  - H La Fe de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Gonzalez-Martin A, Rubio MJ, Heitz F, Depont Christensen R, Colombo N, Van Gorp T, Romeo M, Ray-Coquard I, Gaba L, Leary A, De Sande LM, Lebreton C, Redondo A, Fabbro M, Barretina Ginesta MP, Follana P, Perez-Fidalgo JA, Rodrigues M, Santaballa A, Sabatier R, Bermejo-Perez MJ, Lotz JP, Pardo B, Marquina G, Sanchez-Lorenzo L, Quindos M, Estevez-Garcia P, Guerra Alia E, Manso L, Casado V, Kommoss S, Tognon G, Henry S, Bruchim I, Oaknin A, Selle F. Atezolizumab Combined With Platinum and Maintenance Niraparib for Recurrent Ovarian Cancer With a Platinum-Free Interval >6 Months: ENGOT-OV41/GEICO 69-O/ANITA Phase III Trial. J Clin Oncol. 2024 Dec 20;42(36):4294-4304. doi: 10.1200/JCO.24.00668. Epub 2024 Sep 18. PMID 39292975
- [Derived] Gonzalez Martin A, Sanchez Lorenzo L, Colombo N, dePont Christensen R, Heitz F, Meirovitz M, Selle F, van Gorp T, Alvarez N, Sanchez J, Marques C. A phase III, randomized, double blinded trial of platinum based chemotherapy with or without atezolizumab followed by niraparib maintenance with or without atezolizumab in patients with recurrent ovarian, tubal, or peritoneal cancer and platinum treatment free interval of more than 6 months: ENGOT-Ov41/GEICO 69-O/ANITA Trial. Int J Gynecol Cancer. 2021 Apr;31(4):617-622. doi: 10.1136/ijgc-2020-001633. Epub 2020 Dec 14. PMID 33318079